CLINICAL TRIAL: NCT05194163
Title: A Phase 2a Study of MW150 Stress Kinase Inhibitor in Mild to Moderate Alzheimer's Disease
Brief Title: MW150 Stress Kinase Inhibitor in Mild to Moderate Alzheimer's Disease
Acronym: SKI-AD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neurokine Therapeutics (Industry)
Collaborators: Columbia University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lawrence S Honig, MD, PhD, FAAN, Professor of Neurology at Columbia University Irving Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW150-AD-201; R44AG071388 (NIH)
Record Dates: First submitted 2022-01-13; First posted 2022-01-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease
Keywords: p38alphaMAPK; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — MW01-18-150SRM

STUDY DESIGN:
Intervention Model Description: double-blind randomized placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized through a computerized system by a Data/Statistics Group independent from the investigator or Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10mg MW150 daily (Experimental): 10 mg MW150 daily (1 capsule of 10 mg daily)
  Interventions: Drug: MW150
- placebo daily (Placebo Comparator): placebo daily (1 capsule of matched placebo daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MW150 — oral-delivered capsule of study drug
  Other Names: MW01-18-150SRM
  Arms: 10mg MW150 daily
Drug: Placebo — oral delivered capsule matched to study drug capsule
  Arms: placebo daily

SUMMARY:
This study is a phase 2a randomized double-blind, placebo-controlled, study, in mild-to-moderate Alzheimer's disease, of the oral investigational drug MW150, a p38alphaMAPK kinase inhibitor. The primary goals of this study are to investigate the safety and tolerability, and drug movements in the body. The secondary goals of the study are to investigate the effects of the drug on cognitive performance, activities of daily living, and behavior, and the biological effects of the drug on blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from subject (or legally authorized representative, LAR) and study partner.
2. Male or female, age 50 to 90 inclusive.
3. Have a study partner who is able to accompany the subject, has frequent contact with subject.
4. Meet criteria for Alzheimer's Disease by NIAA-AA criteria.
5. Must speak English fluently.
6. Must have education of at least 8 years.
7. Must have adequate hearing and visual abilities.
8. MMSE score of 14 to 28.
9. Clinical Dementia Rating (CDR) Global score of 0.5 to 2.0 inclusive.
10. Absence of suicidal ideation for at least 1 year.
11. Absence of medical conditions that could affect ability to participate in study.
12. MRI within 1 year of screening, not showing clinically significant structural lesions. Subjects without available MRI within 1 year, must have an MRI performed for eligibility.
13. Stable neuropsychiatric medications for at least 2 months prior to screening.
14. If female, must not be of childbearing potential, as defined by being postmenopausal (more than 1 year without periods) or surgically sterile for at least 6 months prior to screening.
15. If male, must agree to use contraception if with a potentially childbearing partner.

Exclusion Criteria:

1. Presence of clinically significant disorders of the central nervous system other than Alzheimer's disease, such as Lewy Body Disease, Parkinson's disease, hydrocephalus, epilepsy, demyelinating disease, brain tumors, or psychiatric disorders (such as schizophrenia, or severe affective disorders).
2. Serious or unstable hematologic, hepatic, renal, pulmonary, cardiac, or other medical disease.
3. Abnormal liver function tests (ALT or AST) or creatine kinase (CK) upon repeat testing.
4. Chronic hepatitis B or C infection, indicated by positive HBSAg, or HCV-Ab with HCV RNA presence.
5. Known history of human immunodeficiency virus (HIV) infection.
6. Known immune disorder that has a history of requiring treatment with immunosuppressive drugs within the past 1 year.
7. Have a drug or alcohol abuse within 12 months prior to screening.
8. Clinically significant laboratory abnormalities at screening.
9. Screening ECG showing repeated QTcF > 480 msec, or other clinically significant ECG abnormalities.
10. Clinically significant structural brain abnormalities, such as hydrocephalus or intra-axial brain tumors.
11. Participation in another investigational study within 30 days or 5 half-lives prior to screening, whichever is greater.
12. Participation in another study that would have cognitive testing during the duration of this study.
13. History of Covid19 or other viral infections within 3 months.
14. Have a clinically significant medical, surgical, laboratory, or behavioral abnormality, which in the judgment of the Investigator makes the subject unsuitable for the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Drug Safety- Blood tests | 84 days treatment
  Number of participants with treatment-related adverse events as assessed by laboratory test abnormalities.
Drug Safety- Electrocardiographic | 84 days treatment
  Number of participants with emergent abnormal electrocardiograms.
Drug Safety- C-SSRS | 84 days treatment
  Development of any suicidality on COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) score (minimum 0, no maximum, higher number worse).
Drug Tolerability- Adverse events | 84 days treatment
  Incidence of adverse events (AE).

SECONDARY OUTCOMES:
Cognitive change-MMSE | 84 days treatment
  Change in MiniMental State Examination (MMSE) score (0-30, higher score better).
Cognitive change-ADAScog | 84 days treatment
  Change in Alzheimer's Disease Assessment Scale (ADAScog) score (0-70, higher score worse).
Cognitive change-Executive | 84 days treatment
  Change in Trails A (0 - 150 sec) and Trails B test scores (0-300 sec), higher scores worse.
Cognitive change-Language | 84 days treatment
  Change in Verbal Fluency tests for animals and letters (both minimum 0, no maximum, higher scores better).
Functional performance- ADCS-ADL | 84 days treatment
  Change in Alzheimers Disease Cooperative Study Activities of Daily Living (ADCS-ADL) scale (0 - 78, higher score better).
Functional performance-CDR | 84 days treatment
  Change in Clinical Disease Rating Scale (0 - 3, higher score worse).
Behavioral Scale - NPI-Q | 84 days treatment
  Change in Neuropsychiatric Inventory Questionnaire (NPI-Q) (0-36, higher scores worse).
Pharmacodynamics - cytokines | 84 days treatment
  Changes in biomarker measurements of plasma levels of cytokines (IFN-γ, IL-1β, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12P70, IL-22, and TNFα) by Simoa assay (pg/mL).
Pharmacodynamics - neuronal biomarkers | 84 days treatment
  Changes in biomarker measurements of plasma levels of tau protein and NfL protein by Simoa assay (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Honig, MD PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Once study complete, de-identified participant data will be shared upon request by investigators from an academic institution.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: ICF will be shared at onset of enrollment. Study Protocol and SAP will be shared once study published. CSR will be shared once completed.
Access Criteria: Protocol, SAP will be shared via publication. CSR will be shared upon request